CLINICAL TRIAL: NCT05929404
Title: Incidence and Predictors of Bleeding During and Following Endoscopic Retrograde Cholangiopancreatography
Brief Title: Incidence and Predictors of Bleeding During and Following ERCP
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: McGill University (Other); University of Ottawa (Other); Queen's University (Other); Island Health, Victoria, BC (Other); University of Toronto (Other); Radboud University Medical Center (Other); Halton Healthcare (Unknown)
Responsible Party: Sponsor
Other Study IDs: REB 23-0438
Record Dates: First submitted 2023-05-23; First posted 2023-07-03 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Bleeding UGI (During or Post-ERCP)
Keywords: Post-ERCP Bleeding; Intraprocedural Bleeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients on antithrombotic medications: Participants undergoing ERCP procedure taking antithrombotic medications (including antiplatelet and/or anticoagulant medications) at baseline.
- Non-antithrombotic users: Participants undergoing ERCP procedure not taking antithrombotic medications (including antiplatelet and/or anticoagulant medications) at baseline.

SUMMARY:
The incidence of bleeding during ERCP and following ERCP has been estimated using retrospective sources, but granular predictors of bleeding remain unknown, including the use of direct-acting anticoagulants and discontinuation and resumption patterns surrounding their use. In this study, we will aim to assess the incidence and predictors of intra-procedural bleeding during ERCP, and clinically significant post-procedural bleeding following ERCP.

DETAILED DESCRIPTION:
While very effective, endoscopic retrograde cholangiopancreatography (ERCP) is widely known to have the highest adverse event (AE) profile among all commonly performed endoscopic procedures, with a collective AE rate of >10%. Common AEs include post-ERCP pancreatitis, bleeding, cholangitis, cholecystitis, perforation, and cardiopulmonary events. The incidence of bleeding during ERCP and following ERCP has been estimated using retrospective sources, but granular predictors of bleeding remain unknown, including the use of direct-acting anticoagulants and discontinuation and resumption patterns surrounding their use.

It is of critical priority to patients, practitioners, and health administrators to investigate factors associated with all AEs and unplanned healthcare encounters (UHEs) following ERCP, especially given that most ERCPs are performed on an outpatient basis. The per-admission costs of post-ERCP UHEs are substantial. Thus, researchers must prioritize the study of ERCP outcomes, striving to both identify and modify factors leading to AEs and UHEs.

(2) Research Question and Objectives In this study, we will aim to assess the incidence and predictors of intra-procedural bleeding during ERCP, and clinically significant post-procedural bleeding following ERCP.

(3) Methods Design: This is a multicenter prospective cohort study. The primary exposure of interest will be patient use of antithrombotic medications including antiplatelet agents and/or anticoagulant agents. In addition to these variables, other parameters we will assess include: the presence and timing of pharmacologic pancreatitis prophylaxis, extent and timing of trainee involvement, the number and timing of common bile duct (CBD) cannulation attempts, the depth, timing, trajectory and number of pancreatic duct (PD) cannulation(s), the presence and extent of PD opacification, the size(s) of sphincterotomy and/or sphincteroplasty, intra-procedural pathology, and the composition, caliber and length of any PD or CBD stent(s).

Outcomes: The primary outcomes will be clinically significant post-ERCP bleeding (CSPEB), using established definitions, and intra-procedural bleeding, defined as bleeding requiring endoscopic management during ERCP. Secondary outcomes (defined a priori) will include bleeding severity, overall and specific AEs (pancreatitis, cholangitis, cardio-pulmonary events), cannulation time and success rate, as well as overall procedure time and success rate.

Sample Size and Power: Using anticipated CSPEB rates of 2.0% for non-anticoagulant users and 5.0% for anticoagulant users, a minimum of 588 patients in each arm will be required to demonstrate this difference with 80% power and alpha of 0.05.

Statistical Analysis: Variables will be compared using Student's t-test for measured variables and chi-squared test for categorical variables. P values < 0.05 will be considered significant. We will use multivariable logistic regression to assess associations between risk factors and having bleeding versus not having bleeding. Clinically relevant subgroup analyses will also be performed by relevant patient-, endoscopist-, and procedure-related characteristics. Odds ratios per outcome will be reported with 95% CIs.

ELIGIBILITY:
Inclusion Criteria:

* Subject referred for ERCP, regardless of indication;
* Subject age 18 years or older;
* Subject able to give informed consent to involvement be included.

Exclusion Criteria:

* Subject has a standard contraindication to ERCP;
* Subject or surrogate unable or unwilling to provide informed consent;
* Subject age < 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to a hospital-based endoscopy unit for consideration of ERCP.
Sampling Method: Non-Probability Sample
Enrollment: 5872 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Clinically significant post-ERCP bleeding | 30 days
  Clinically significant post-ERCP bleeding will be defined using established definitions (Cotton et al. Gastrointest Endoscopy 2010; Forbes et al. Gut 2022).

CONTACTS AND LOCATIONS:
Overall Officials: Nauzer Forbes, MD MSc, Principal Investigator — Peter Lougheed Center
Locations (1):
- Peter Lougheed Center, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Bishay K, Ruan Y, Barkun AN, Chen YI, Singh A, Hookey L, Arya N, Calo NC, Grover SC, Siersema PD, Thosani N, Darvish-Kazem S, Siegal D, Bass S, Cole M, Lei Y, Li S, Mohamed R, Turbide C, Chau M, Howarth M, Cartwright S, Koury HF, Nashad T, Meng ZW, Tepox-Padron A, Kayal A, Gonzalez-Moreno E, Brenner DR, Smith ZL, Keswani RN, Elmunzer BJ, Wani S, Bridges RJ, Hilsden RJ, Heitman SJ, Forbes N. Incidence, Predictors, and Outcomes of Clinically Significant Post-Endoscopic Retrograde Cholangiopancreatography Bleeding: A Contemporary Multicenter Study. Am J Gastroenterol. 2024 Nov 1;119(11):2317-2325. doi: 10.14309/ajg.0000000000002946. Epub 2024 Jul 5. PMID 39495582